CLINICAL TRIAL: NCT02726243
Title: Intestinal Microbiota and Colorectal Cancer in Inflammatory Bowel Disease - DYSCOLIC
Brief Title: Intestinal Microbiota and Colorectal Cancer in Inflammatory Bowel Disease
Acronym: DYSCOLIC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: NI13006
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Inflammatory Bowel Disease; Colorectal Cancer
Keywords: Inflammatory bowel disease; Crohn's Disease; Ulcerative Colitis; colorectal cancer; primary sclerosing cholangitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colorectal Neoplasms; Crohn Disease; Colitis, Ulcerative; Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stools
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- IBD without CRC
- IBD with CRC
- IBD with dysplasia
- non IBD without CRC
- non IBD with CRC
- IBD-PSC without CRC
- IBD-PSC with CRC
- IBD-PSC with dysplasia or healthy subjects: IBD-PSC with dysplasia or healthy subjects for whom a colonoscopy is scheduled

SUMMARY:
Build a collection of fecal microbiota in order to determine the characteristics of gut microbiota associated with colorectal cancer in Inflammatory bowel disease (IBD).

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) are chronic and relapsing disabling disease. Crohn's disease (CD) and Ulcerative colitis (UC) are the two main types of IBD.

Patients with IBD are at greater risk of intestinal infection including viral infections (including cytomegalovirus) and bacterial (especially Clostridium difficile). In the long term, patients with colonic involvement are at an increased risk of colorectal cancer (CRC). Moreover, it has been reported in several cohort studies that patients with primary sclerosing cholangitis (PSC) associated with IBD (PSC-IBD), have an even increased risk of CRC (about 10 to 20% at 10 years). Other studies also suggest that the microbiota has an impact on liver diseases. Conversely, cholestatic liver diseases (such as PSC) can influence the microbiota, notably through modification of the production of bile acids. Finally, the role of the gut microbiota in the development of the CRC in IBD has been well established in animal models. The pathophysiological mechanisms are not well understood but may involve an alteration of the balance between protective bacteria against harmful microbiota.

This study aims to investigate the link between gut microbiota, intestinal inflammation, colorectal cancer, bile acid and liver diseases and this, through the creation of a biological collection of fecal microbiota from fecal samples from 8 groups of subjects: (i) IBD without CCR (ii) IBD with CCR, (iii) IBD with dysplasia, (iv) non IBD without CCR, (v) non IBD with CCR, (vi) IBD-CSP without CCR, (vii ) IBD-CSP with CCR, (viii) IBD-CSP with dysplasia. In these patients, microbiota composition will be assessed by sequencing technology.

ELIGIBILITY:
Inclusion Criteria:

* Patient with the capacity to give informed consent.
* Age ≥ 18 years.
* A patient with IBD (Crohn's disease or ulcerative colitis) or healthy subject having a screening colonoscopy scheduled.
* Diagnosis of pathologies in question established or confirmed in any of the services involved in the study and according to international diagnostic criteria (Consensus ECCO).
* Patient follow-up in one of the services involved in the study

Exclusion Criteria:

* trusteeship, guardianship or safeguard justice.
* Subject does not speak French.
* Subject unable to answer questions or to speak.
* Previous history of colonic resection
* Taking antibiotics within 8 weeks preceding the stool sample Temporary exclusion criterium)
* Taking a bowel preparation for colonoscopy within 6 weeks before the stool sample (temporary exclusion criterium). Sampling is possible before bowel preparation or on the first stool after starting the bowel preparation.
* Ostomy at the time of sampling
* Current treatment by radiotherapy, chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with or without an inflammatory bowel disease, for whom a colonoscopy is scheduled.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2014-11; Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Composition of fecal microbiota by 16S sequencing | Baseline
  Microbiota composition will be assessed using MiSeq technology

SECONDARY OUTCOMES:
Profile of fecal bile acids | Baseline
  Characterize the profile of fecal bile acids of the patients included in the biological. collection. After extraction, the bile acid profile will be determined by LC-MS / MS (liquid chromatography coupled to tandem mass spectrometry).
  - Characterize some cultivable species of gut microbiota of patients included in the study by culture. Aerobic and anaerobic bacterial strains will be isolated from patients stools and stored for further characterization.

CONTACTS AND LOCATIONS:
Overall Officials: Harry SOKOL, MD PhD, Principal Investigator — APHP
Locations (1):
- Gastroenterology Department of Saint Antoine Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lavelle A, Nancey S, Reimund JM, Laharie D, Marteau P, Treton X, Allez M, Roblin X, Malamut G, Oeuvray C, Rolhion N, Dray X, Rainteau D, Lamaziere A, Gauliard E, Kirchgesner J, Beaugerie L, Seksik P, Peyrin-Biroulet L, Sokol H. Fecal microbiota and bile acids in IBD patients undergoing screening for colorectal cancer. Gut Microbes. 2022 Jan-Dec;14(1):2078620. doi: 10.1080/19490976.2022.2078620. PMID 35638103